CLINICAL TRIAL: NCT04188262
Title: Natural Vascular Scaffolding (NVS) Therapy for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA)
Brief Title: Natural Vascular Scaffold (NVS) Therapy for Treatment of Atherosclerotic Lesions (Activate I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alucent Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1060-002
Record Dates: First submitted 2019-12-04; First posted 2019-12-05 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Catheterization, Peripheral
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: NVS Therapy will be delivered to de novo lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) during PTA in patients with symptomatic peripheral artery disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NVS Therapy (Experimental): NVS Therapy will be delivered to de novo lesions in Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) during PTA in patients with symptomatic peripheral artery disease.
  Interventions: Combination Product: NVS Therapy

INTERVENTIONS:
Combination Product: NVS Therapy — Combination Product: NVS Therapy which includes NVS Injection (investigational product) and the following investigational devices: NVS Delivery Catheter, NVS light Fiber, and NVS light source.
  Other Names: Natural Vascular Scaffold

SUMMARY:
The NVS Therapy is being studied to evaluate the safety and efficacy to facilitate retention of acute luminal gain, leading to acute hemodynamic improvement in superficial femoral and popliteal arteries with reference vessel diameters between 4.0 and 7.0 mm and lesion lengths less than or equal to 56mm.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center, open label Phase 1 study to assess the safety, pharmacokinetics (PK), and preliminary efficacy trends to applying NVS therapy to de novo lesions in the superficial femoral artery (SFA) and the proximal popliteal artery (PPA) during percutaneous transluminal angioplasty (PTA) in patients with life-style limiting claudication due to obstructive SFA and proximal popliteal artery atherosclerosis. Each investigator will receive supervised training for each procedure.

Eligibility to participate in the study is determined during the screening period and prior to the index procedure with the NVS therapy. Study Data will be analyzed through the Day 365 follow-up visit.

ELIGIBILITY:
General Description of Subject Population: Adults with symptoms of claudication and/or rest pain (Rutherford Classification 2, 3, or 4) (see Appendix 3) and angiographic evidence of an atherosclerotic lesion of the superficial femoral artery and/or proximal popliteal artery ≥70% diameter stenosis and < 100% stenosis.

Subjects must meet all of the following general eligibility criteria:

1. Subject is at least 18 years of age.
2. Subject (or legally authorized representative [LAR]) understands the study requirements and the treatment procedure and provides written informed consent before any study-specific tests or procedures are performed.
3. Subject is eligible for PTA.
4. Subject is willing to comply with all protocol required follow-up evaluations.
5. Subject has documented Rutherford Classification 2 to 4 (see Appendix 3).
6. Subject has laboratory test results that are within clinically acceptable limits.
7. In investigator's opinion, subject is hemodynamically stable at the time of the index procedure.
8. Subject has a life expectancy of ≥ 1 year in the opinion of the Investigator.
9. Subject is able to tolerate the insertion of a 7F sheath into the common femoral artery (CFA), as determined by the investigator.
10. Subject is able to undergo contralateral access, as determined by the Investigator.

Exclusion Criteria:

Subjects must not meet any of the following general eligibility criteria:

1. Subject had cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 3 months prior to enrollment with any residual deficit involving the index lower extremity.
2. Subject has any permanent neurologic defect that may impair ambulation and/or cause non-compliance with the protocol.
3. Subject had a STEMI or NSTEMI within the last 3 months prior to enrollment.
4. Subject is pregnant, breastfeeding, or planning to become pregnant in the next 365 days. Subjects (male and female) must agree to use effective birth control measures for duration of study.
5. Subject is currently receiving oral or intravenous immunosuppressive therapy (e.g., inhaled steroids are not excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Freedom from all-cause mortality, freedom from target limb major amputation, freedom from target lesion revascularization (TLR). | Day 30
  The overall composite occurrence of participants free from all-cause mortality, target limb major amputation, target lesion revascularization (TLR) through post-index procedure Day 30 will be summarized as a percentage.
NVS Drug Plasma Concentrations | Day 1 - 24 (Or Discharge)
  The Peak Plasma Concentration (Cmax) will be determined from plasma 10-8-10 Dimer concentrations for blood samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hauser, Study Director — Alucent Biomedical
Locations (4):
- United States (4):
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Mid-Michigan Heart & Vascular Center, Saginaw, Michigan
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: No